CLINICAL TRIAL: NCT05939739
Title: Study of the Value of Trio Exome Sequencing in the Etiological Assessment of Specific Non-syndromic Language and Learning Disorders
Acronym: TSLA ES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DELANNE PHRCI 2021
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Specific Language and Learning Disorders (SLLD)
MeSH Terms: conditions — Learning Disabilities | interventions — Blood Specimen Collection; Referral and Consultation; Social Sciences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood samples — Samples collected during blood sampling for array CGH (1 EDTA tube for index case and 2 biological relatives)
Other: Consultation for results delivery — at 4 months
Other: Study Humanities and Social Sciences — Interview offered to 20 families with positive results and 10 families with negative results

SUMMARY:
Specific language and learning disorders (SLLD) affect around 5-10% of school-aged children, or 1-2 child(ren) per class. SLLDs correspond to the impairment of a specific cognitive function and are divided into 5 categories: dyslexia, dysphasia, dyspraxia, dyscalculia and attention deficit hyperactivity disorder (ADHD) (DSM-5). In recent years, real progress has been made in their clinical diagnosis and management, thanks to a better description of these disorders in the DSM-5 and the advent of rehabilitative treatments (neuropsychology, speech therapy, occupational therapy, orthoptics, etc.). SLLD can occur in a sporadic or familial context (sibling involvement, a symptomatic parent, other relatives who may mimic dominant inheritance with variable expressivity and incomplete penetrance).

It has long been suspected that SLLD is secondary to multifactorial inheritance, with a combination of frequent genetic variations and environmental factors. In France, in the absence of an obvious syndromic diagnosis, the current strategy is to prescribe array CGH, combined in girls with a search for fragile X syndrome (in boys, this syndrome leads to systematic intellectual disability, which does not justify its study in SLLD). A few genes have been described as being specifically involved in a small proportion of SLLD, most often with de novo variations or inherited from a symptomatic parent. There are no distinctive clinical features to guide targeted sequencing of these genes. Moreover, our recent experience shows that genes implicated in intellectual disability may also be involved in SLLD. Very few studies have been published in the literature evaluating the value of exome sequencing in SLLD. Only two studies have been identified, involving 10 and 43 patients with specific SLLD.

In view of the roll-out of the French Genomic Medicine Plan (PFMG 2025), it is important to set up a study aimed at assessing the value of genome-wide sequencing in the etiological work-up for SLLD.

Participation in the study consists of:

* an inclusion visit, where an additional blood sample will be taken during the baseline work-up
* a results visit (4 months after the inclusion visit)

Optional qualitative study: semi-structured interview 1 year after the inclusion visit proposed to 20 patients or families with a positive result and to 10 patients with a negative result.

ELIGIBILITY:
Inclusion Criteria:

* Index case suffering from one or more severe learning disorders (requiring in-school help or intensive rehabilitation), justified by neuropsychological and/or speech therapy and/or occupational therapy assessments, reviewed by experts and supplemented if necessary within the framework of the study, and not yet having undergone genetic testing.
* Index case aged 3 to 40 years
* Sample may be taken from index case and 2 known biological parents
* Consent signed by the parents and by the index case if major
* Index case and parents covered by national health insurance

Exclusion Criteria:

* Index case and parents have a condition which, in the opinion of the investigator, would contraindicate the subject's participation in the study.
* Intellectual disability confirmed by neuropsychological testing or strongly suspected clinically in the index case and/or his/her parents
* Obvious syndromic diagnosis (syndrome or antecedents having definitely led to a developmental disorder)
* Persons deprived of liberty by judicial or administrative decision,
* Adults under guardianship,
* Persons residing in a health or social establishment
* Patients in critical situations
* Pregnant, parturient or nursing women
* Previous array CGH and/or Fragile X testing or any other targeted genetic examination (except standard karyotype).

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Identification of a genetic cause defined by the presence of at least one ACMG class 4 or 5 variant. | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No